CLINICAL TRIAL: NCT07076134
Title: A Pilot Trial of a Community-and Primary Care-based Intervention Linked With mObile Technology for Hypertension Control in Nepal (CoPILOT Trial)
Brief Title: Community-and Primary Care-based Intervention Linked With mObile Technology for HTN Control in Nepal
Acronym: CoPILOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke Kunshan University (Other)
Collaborators: Dhulikhel Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 437_2024; DGHI pilot grant (Other Grant/Funding Number: Duke Global Health Institute)
Record Dates: First submitted 2024-11-19; First posted 2025-07-21 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): FCHVs and FLHWs will be given 2 days training on Android mobile-based application usage. The app includes prompts regarding patients' current BP measurements and educational content on dietary habits, the importance of physical activity, and the harmful effects of smoking and alcohol consumption. FCHVs will conduct bimonthly meetings with groups of hypertensive patients. They will measure BP, enter it in the app, provide awareness and refer to nearby health facilities if needed. Data entered by FCHVs will be synchronized with FLHWs' accounts, allowing them to view the data entered by FCHVs. After a patient visits a health facility, the FLHW will take action as needed and record it in the app, thereby creating a linkage between the community and the health facility. Patients registered in the app will also receive weekly health education text messages on their mobile phones.
  Interventions: Other: FCHVs and FLHWs in a community managing HTN using primary care based approach and mobile health technology
- Usual care (No Intervention): Usual care refers to the standard treatment that participants receive as part of their regular routine, without the research introducing any new interventions. The FCHVs and FLHWs in the usual care group will not receive training on application usage, and the participants will not receive text messages on their mobile phones.

INTERVENTIONS:
Other: FCHVs and FLHWs in a community managing HTN using primary care based approach and mobile health technology — Our intervention utilizes FCHVs as a bridge between the community and health facilities to improve HTN care. FCHVs and FLHWs will receive 2 days of training to use an Android app. The app provides prompts for BP measurement and educational content on healthy lifestyles. For 3 months, FCHVs will conduct bimonthly meetings, measure BP, height, and weight, provide awareness and enter sociodemographic details of participants into the app. Participants with BP ≥130/85 mmHg (unmedicated) or ≥120/80 mmHg (on medication) will be referred to a nearby health facility by FCHVs. The data entered by FCHVs will be linked to FLHWs' terminals. FLHWs will enter required information about medication use, referrals, and follow-ups into the app and take necessary actions for the treatment of referred patients. The intervention includes 795 participants from 10 clusters with BP ≥130/85 mmHg. Data on BP, medication adherence, quality of life, and physical activity will be collected at baseline and endline.
  Arms: Intervention group

SUMMARY:
The clinical trial aims to evaluate whether a community and primary care-based intervention linked with mobile technology (CoPILOT) is acceptable, effective, cost-effective, sustainable, and scalable in improving hypertension (HTN) control among individuals aged 30 to 70 in Nepal. The primary research questions include:

Is the use of the application by Frontline Health Workers (FLHWs) and Female Community Health Volunteers (FCHVs) feasible and acceptable? Can FCHVs equipped with mHealth technology effectively increase the linkage of individuals with elevated blood pressure (BP) to health facilities? Does a mobile-based lifestyle intervention reduce or control BP? Can adherence to prescribed HTN treatments be improved among patients through this intervention?

DETAILED DESCRIPTION:
The researcher will compare the intervention and control groups to assess changes in BP, quality of life (QoL), body mass index (BMI), medication adherence, and linkage to care.

Participants in the intervention group will:

Attend bi-monthly meetings conducted by FCHVs for BP measurement, facilitated through the mobile application.

Receive healthy lifestyle awareness guidance provided by FCHVs via the mobile app and supplemented with text message reminders.

Visit nearby health facilities for monthly follow up.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patient's should be in the range of 30 to 70 years old living in selected communities with HTN (systolic BP ≥ 130 mmHg or diastolic ≥ 85 mmHg or taking antihypertensive medication)
* They should have been diagnosed previously and under medication.
* They should agree to the informed consent
* FCHVs should be working for the selected communities and agree to the informed consent
* FLHWs should work for the health facilities in selected communities and agree to the informed consent.

Exclusion Criteria:

* Participants who are not able to respond during the data collection period.
* Participants who are out of municipality during the data collection period.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure (mmHg) | Three months intervention
  Change in systolic and diastolic blood pressure (mmHg) among hypertensive patients in the intervention group will be measured using a validated digital blood pressure monitor at baseline and endline. The outcome will be reported as the mean change in systolic and diastolic blood pressure.

SECONDARY OUTCOMES:
Change in body weight(kg) | During baseline and endline (3 months intervention period)
  Weight will be measured in kilograms using a weighing scale at health posts by healthcare providers or by FCHVs during group meetings. The measurements will be recorded in the application and later analyzed to assess changes in body weight.
Height (meters) | At baseline or endline (3 months intervention period)
  FLHWs will measure the height (in meters) by using stadiometer at health posts. They will enter the data in the application.
Change in body mass index (BMI) (kg/m²) | Three months intervention period
  Body Mass Index (BMI) will be calculated using the formula BMI = weight (kg) / height² (m²). The BMI values will be derived from the collected data and analyzed to assess changes.
Change in quality of life as measured by EuroQol Visual Analogue Scale (EQ VAS) | Three months intervention period
  Quality of life will be assessed using the EuroQol Visual Analogue Scale (EQ VAS), administered by the study team at baseline and endline. Participants will rate their overall health on a vertical visual analogue scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state), and changes in these scores will be used to evaluate improvements in health-related quality of life.
Change in antihypertensive medication adherence as measured by the Morisky Green Levine Medication Adherence Scale (MGLS) | Three months intervention period
  Medication adherence will be assessed using the Morisky Green Levine Medication Adherence Scale (MGLS), administered by the study team at baseline and endline. The MGLS is a 4-item self-report scale that assesses medication-taking behavior, with each item scored 1 for "No" and 0 for "Yes." Total scores range from 0 to 4, with higher scores indicating better adherence. The outcome will be reported as the change in MGLS total score over the 3-month intervention period.
Change in perceived empowerment among FCHVs and FLHWs as assessed through structured qualitative interviews | Three months intervention period
  Empowerment will be assessed through qualitative semi-structured interviews conducted with FCHVs and FLHWs at both baseline and endline. Interview questions will explore changes in core dimensions of empowerment, including knowledge, confidence, and role perception, in relation to the hypertension mHealth intervention. Interviews will be audio-recorded, transcribed verbatim, and analyzed using thematic analysis. The outcome will be reported as a summary of key themes and illustrative quotes that reflect perceived changes in empowerment over the 3-month intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Namobuddha municipality, Namobuddha, Kavrepalanchowk, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He J, Irazola V, Mills KT, Poggio R, Beratarrechea A, Dolan J, Chen CS, Gibbons L, Krousel-Wood M, Bazzano LA, Nejamis A, Gulayin P, Santero M, Augustovski F, Chen J, Rubinstein A; HCPIA Investigators. Effect of a Community Health Worker-Led Multicomponent Intervention on Blood Pressure Control in Low-Income Patients in Argentina: A Randomized Clinical Trial. JAMA. 2017 Sep 19;318(11):1016-1025. doi: 10.1001/jama.2017.11358. PMID 28975305
- [Background] Lloyd-Sherlock P, Beard J, Minicuci N, Ebrahim S, Chatterji S. Hypertension among older adults in low- and middle-income countries: prevalence, awareness and control. Int J Epidemiol. 2014 Feb;43(1):116-28. doi: 10.1093/ije/dyt215. Epub 2014 Feb 6. PMID 24505082
- [Background] Tian M, Ajay VS, Dunzhu D, Hameed SS, Li X, Liu Z, Li C, Chen H, Cho K, Li R, Zhao X, Jindal D, Rawal I, Ali MK, Peterson ED, Ji J, Amarchand R, Krishnan A, Tandon N, Xu LQ, Wu Y, Prabhakaran D, Yan LL. A Cluster-Randomized, Controlled Trial of a Simplified Multifaceted Management Program for Individuals at High Cardiovascular Risk (SimCard Trial) in Rural Tibet, China, and Haryana, India. Circulation. 2015 Sep 1;132(9):815-24. doi: 10.1161/CIRCULATIONAHA.115.015373. Epub 2015 Jul 17. PMID 26187183
- [Background] Yan LL, Gong E, Gu W, Turner EL, Gallis JA, Zhou Y, Li Z, McCormack KE, Xu LQ, Bettger JP, Tang S, Wang Y, Oldenburg B. Effectiveness of a primary care-based integrated mobile health intervention for stroke management in rural China (SINEMA): A cluster-randomized controlled trial. PLoS Med. 2021 Apr 28;18(4):e1003582. doi: 10.1371/journal.pmed.1003582. eCollection 2021 Apr. PMID 33909607
- [Background] Ni Z, Atluri N, Shaw RJ, Tan J, Khan K, Merk H, Ge Y, Shrestha S, Shrestha A, Vasudevan L, Karmacharya B, Yan LL. Evaluating the Feasibility and Acceptability of a Mobile Health-Based Female Community Health Volunteer Program for Hypertension Control in Rural Nepal: Cross-Sectional Study. JMIR Mhealth Uhealth. 2020 Mar 9;8(3):e15419. doi: 10.2196/15419. PMID 32149712
- [Background] Tan J, Xu H, Fan Q, Neely O, Doma R, Gundi R, Shrestha B, Shrestha A, Shrestha S, Karmacharya B, Gu W, Ostbye T, Yan LL. Hypertension Care Coordination and Feasibility of Involving Female Community Health Volunteers in Hypertension Management in Kavre District, Nepal: A Qualitative Study. Glob Heart. 2020 Oct 23;15(1):73. doi: 10.5334/gh.872. PMID 33150138
- [Background] Bhattarai P, Shrestha A, Xiong S, Peoples N, Ramakrishnan C, Shrestha S, Yin R, Karmacharya B, Yan LL, Jafar TH. Strengthening urban primary healthcare service delivery using electronic health technologies: A qualitative study in urban Nepal. Digit Health. 2022 Jul 21;8:20552076221114182. doi: 10.1177/20552076221114182. eCollection 2022 Jan-Dec. PMID 35898291
- See also: The WHO Nepal launched the Hypertension Care Cascade Initiative on May 17, 2023, aiming to improve hypertension prevention and treatment across the country. This initiative focuses on strengthening healthcare systems and enhancing community-based care — https://www.who.int/nepal/news/detail/17-05-2023-hypertension-care-cascade-initiative-launched
- See also: The clinical trial NCT06163859 focuses on evaluating the effectiveness of a new intervention for managing hypertension. The study aims to improve patient outcomes and refine treatment strategies — https://clinicaltrials.gov/study/NCT06163859